CLINICAL TRIAL: NCT04441931
Title: A Phase 1, Randomized, Placebo-Controlled Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Immunogenicity of LY3832479 Given as a Single Intravenous Dose in Healthy Participants
Brief Title: A Study of LY3832479 (LY-CoV016) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 18029; J2Z-MC-PGAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — etesevimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3832479 (Experimental): Participants received single Intravenous (IV) doses of 700, 2800 and 7000 milligrams (mg) LY3832479.
  Interventions: Drug: LY3832479
- Placebo (Placebo Comparator): Participants received single IV dose of Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3832479 — Administered IV.
  Other Names: LY-CoV016
  Arms: LY3832479
Drug: Placebo — Administered IV.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about the safety of LY3832479 and any side effects that might be associated with it. Blood tests will be done to measure how much LY3832479 is in the bloodstream and how long it takes the body to eliminate it. Participation could last up to 16 weeks and may include up to 10 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history and physical examination

Exclusion Criteria:

* Test positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
* Pregnant women and women of childbearing potential
* Have a history or presence of cardiovascular (including hypertension), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders that, in the opinion of the investigator, are capable of significantly altering the absorption, metabolism, or elimination of drugs, or of constituting a risk while taking the investigational product, or of interfering with the interpretation of data
* Have participated in a clinical study involving an investigational product, with last dose within the past 30 days or 5 half-lives (whichever is longer) prior to dosing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- Pooled Placebo: Participants received single Intravenous (IV) dose of Placebo.
- 700 mg LY3832479 IV: Participants received single IV dose of 700 mg LY3832479.
- 2800 mg LY3832479 IV: Participants received single IV dose of 2800 mg LY3832479.
- 7000 mg LY3832479 IV: Participants received single IV dose of 7000 mg LY3832479.
Period: Overall Study
Arm/Group | Pooled Placebo | 700 mg LY3832479 IV | 2800 mg LY3832479 IV | 7000 mg LY3832479 IV
Started | 6 | 7 | 7 | 6
Received at Least One Dose of Study Drug | 6 | 7 | 7 | 6
Completed | 6 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | 700 mg LY3832479 IV | 2800 mg LY3832479 IV | 7000 mg LY3832479 IV | Total
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (10.8) | 41.0 (7.4) | 41.4 (11.2) | 45.7 (8.9) | 42.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 0 | 3
  Male | 5 | 6 | 6 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5 | 1 | 11
  Not Hispanic or Latino | 3 | 5 | 2 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 0 | 1 | 7
  White | 1 | 5 | 6 | 4 | 16
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 | 7 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug
Description: The number of participants with 1 or more SAEs assessed as related to the study drug and is summarized cumulatively. A serious adverse event is defined as an event that results in death, initial or prolonged hospitalization, is life-threatening, leads to persistent or significant disability/incapacity, is associated with congenital anomaly/birth defect, or is considered significant by the investigator for any other reason. A summary of all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through Follow-up (Week 12)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Pooled Placebo | 700 mg LY3832479 IV | 2800 mg LY3832479 IV | 7000 mg LY3832479 IV
Number analyzed (Participants) | 6 | 7 | 7 | 6
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time 0 to Infinity (AUC[0-∞]) of LY3832479
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time 0 to infinity (AUC[0-∞]) of LY3832479.
Time Frame: Day 1 (predose, end of infusion, 6 hours after start of infusion), 2, 3, 8, 15, 29, 43, 57, 85
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day per milliliter(ug*day/mL)
Arm/Group | 700 mg LY3832479 IV | 2800 mg LY3832479 IV | 7000 mg LY3832479 IV
Number analyzed (Participants) | 7 | 7 | 6
micrograms*day per milliliter(ug*day/mL) | 4920 (23) | 22700 (22) | 50800 (33)

3. Secondary Outcome: PK: Maximum Serum Concentration (Cmax) of LY3832479
Description: PK: Maximum Serum Concentration (Cmax) of LY3832479.
Time Frame: Day 1 (predose, end of infusion, 6 hours after start of infusion), 2, 3, 8, 15, 29, 43, 57, 85
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | 700 mg LY3832479 IV | 2800 mg LY3832479 IV | 7000 mg LY3832479 IV
Number analyzed (Participants) | 7 | 7 | 6
ug/mL | 244 (24) | 1130 (14) | 2390 (23)

ADVERSE EVENTS:
Time Frame: Baseline, upto 3 Months
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Pooled Placebo IV: Participants received single Intravenous (IV) dose of Placebo.
Arm/Group | Pooled Placebo IV | 700 mg LY3832479 IV | 2800 mg LY3832479 IV | 7000 mg LY3832479 IV
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 2/7 | 2/7 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo IV (N=6) | 700 mg LY3832479 IV (N=7) | 2800 mg LY3832479 IV (N=7) | 7000 mg LY3832479 IV (N=6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT04441931/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT04441931/SAP_001.pdf